CLINICAL TRIAL: NCT00710723
Title: Vitrification Versus Slow Freezing of Human Day 3 Embryos
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Gasthuisberg (Other)
Responsible Party: Prof. Dr. Thomas D'Hooghe, University Hospital, Gasthuisberg.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: dwille1
Record Dates: First submitted 2008-01-04; First posted 2008-07-04 (Estimated); Last update posted 2008-07-04 (Estimated); Status verified 2008-01

CONDITIONS: Cleavage Stage, Ovum
MeSH Terms: interventions — Vitrification

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- 1 (Experimental): vitrification
  Interventions: Procedure: vitrification
- 2 (No Intervention): Slow freezing

INTERVENTIONS:
Procedure: vitrification — Vitrification using Hemi-straw carrier system.
  Arms: 1

SUMMARY:
In assisted reproduction technology (ART), cryopreservation of embryos maximizes the potential of IVF cycles. Currently different cryopreservation methods are used, the conventional slow freezing method and vitrification. There is, therefore an immediate need to assess which cryopreservation technique is preferential in human IVF. In this prospective randomised study conventional slow freezing and vitrification, using the Hemi-straw carrier system, of human day 3 embryos were compared.

DETAILED DESCRIPTION:
1. Background

   Although there are studies that reported successful pregnancies after transfer of vitrified cleavage stage embryos, most of the studies focused on the vitrification of oocytes and blastocysts. As far as we know, there is only one report of a randomised prospective study were both common freezing methods -conventional slow freezing and vitrification (making use of the nylon loop system with 40% ethylene glycol), were compared for day 3 embryos (Rama Raju, Haranath et al., 2005). They report an implantation and pregnancy rate (14,9% and 35,0% respectively) with vitrification, which is significantly higher than the rates with the slow freezing protocol (4,2% and 17,4% respectively). There is still need to more randomised studies which compares both freezing methods for cleavage stage embryos .

   There is evidence in literature that the vitrification method used at LUFc (hemi-straw) is superior to the method used in the randomised trial of Rama Raju. Liebermann and Tucker compared both the hemi-straw and cryoloop system for vitrification of day 3 embryos derived from abnormally fertilized zygotes (Liebermann and Tucker, 2002). They found no statistical difference (p=0.07) in the survival rate, but the development after 24 hours was statistically better (p =0.002) using hemi-straws. Based on this study we would even expect better results than the study of Rama Raju.

   To further refine the effect of cryopreservation of cleavage stage embryos using the hemi-straw system on developmental and implantation potential, the effectiveness of vitrification (20% EG and 20% DMSO) was compared with slow freezing.
2. Materials and methods

   * Patients In this prospective study all patients underwent IVF or ICSI between are included. Fresh embryo transfer was carried out on day 3 after insemination. All surplus embryos who reached at least the 6 cell stage on day 3 and had less than 20% fragmentation were considered for cryopreservation using either vitrification or slow freezing.
   * Randomisation All embryos will be cryopreserved by one of the two methods. Randomisation will take place at day 3 after insemination. For practical reasons, all embryos frozen on the same day will be randomly assigned to the same freezing method.
   * Results from retrospective data analysis Vitrification has been used as a standard cryopreservation method at the LUFc since September 2004. So both slow freezing and vitrification had been used for cryopreservation of day 3 embryos. The method used depends on workload… so there was no randomisation. After a retrospective analysis of these data (124 cycles 43 in the slow group and 81 in the vitrification group), we noticed a significant increase in the survival of the embryos after vitrification (81.2% in the vitrification group versus 45.8% in the slow group; p<0.0001). There was no significant difference in pregnancy rate between both groups (19.8% in the vitrification versus 30.2% in slow group; p=NS).

   So far we saw a remarkable difference in survival immediately or 24h after thawing, but a clear difference in the implantation rate has not been discovered yet, therefore we would like to start a randomised trial to proof a significant difference at the implantation or pregnancy level.
   * Vitrification of human embryos Our method was based on the procedure described by Vanderzwalmen et al 2000 (Vanderzwalmen, Bertin et al., 2000). First the embryos were equilibrated (PBS with 17% HSA ) for 2 min at room temperature. They were then transferred to the first vitrification solution (PBS + 14% HSA + 10% DMSO + 10% ethylene glycol) for 2 min at RT followed by 30 sec in the second vitrification solution (PBS + 12% HSA + 20 % DMSO + 20% ethylene glycol + ficoll + sucrose). Finally the embryos were loaded as quickly as possible on the Hemi-straw in a droplet of approximately 3 µl and immersed directly in liquid nitrogen. Afterwards the hemi-straw was inserted in the CBS-straw.
   * Thawing after vitrification The hemi-straw holding exactly one embryo was pulled out of the CBS straw and immediately immersed into 3 ml of the first thawing solution (PBS with 20% HSA) for 3 min at 36°C. Afterwards the embryo was consecutively exposed for 2 min to the 3 other thawing solutions (0.5M sucrose, 0.25M sucrose and 0.125M sucrose respectively). The embryos were washed thoroughly and incubated overnight in COOK blastocyst medium. Embryos are considered as 'survived' if at least 50% of the blastomeres survived the vitrification procedure.
   * Slow freezing and thawing procedure For the slow freezing and thawing procedure we used the HEPES-buffered commercial freezing medium of Cook (K-SICS 5000) with propandiol and sucrose as cryoprotectants.
3. Statistical analysis and power calculation

Based on literature (Rama Raju et al 2005) we expect a 10 % higher implantation rate in the vitrification group (25%) versus the slow freezing group (15%)(Rama Raju, Haranath et al., 2005). To proof a significant difference at the implantation or pregnancy level with α=0,05 and a power (β) of 0,80. Therefore we would need 270 embryos transferred in each group.

ELIGIBILITY:
Inclusion Criteria:

* Embryos of sufficient embryo quality: at least 6 cells on day 3 and less than 20 % fragmentation.

Ages: 18 Years to 43 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 901 (Actual)
Dates: Start 2005-10; Study Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy rate | 9 months

SECONDARY OUTCOMES:
survival rate after thawing of embryos | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: D'Hooghe Thomas, Prof. Dr., Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium